CLINICAL TRIAL: NCT00395356
Title: Efficacy and Feasibility of an Intermittent Weight Loss Program: A Pilot Study.
Brief Title: Efficacy and Feasibility of an Intermittent Weight Loss Program.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FRSQ-5574
Record Dates: First submitted 2006-11-01; First posted 2006-11-02 (Estimated); Last update posted 2006-11-02 (Estimated); Status verified 2006-11

CONDITIONS: Obesity
Keywords: Diet; Caloric restriction; Intermittent diet; Obesity; Postmenopausal women
MeSH Terms: conditions — Obesity | interventions — Caloric Restriction

INTERVENTIONS:
Behavioral: calorie controlled diet

SUMMARY:
The goal of the study is to measure the effect of an approach including phases of active weight loss broken by weight stabilisation periods (named intermittent weight loss) on the metabolic profile.

First, the intermittent weight loss approach will contribute to create an artificial transitory steady state during the weight loss treatment that will help to minimize the adverse effects of the standard approach on muscle mass and resting metabolic rate. Second, despite a comparable fat mass loss, the intermittent weight loss approach will improve the metabolic profile to a greater degree compared to the standard approach. Finally, the intermittent weight loss approach will be associated with less weight regain after the treatment since the beneficial effect on muscle mass and metabolic rate.

DETAILED DESCRIPTION:
Excessive levels of body fat are associated with metabolic disturbances predictive of an increased risk of coronary heart disease (CAD). It is presently unclear as to the magnitude of weight loss needed to accrue metabolic benefits. Despite the effectiveness of weight loss to reduce obesity levels, studies have shown that only minor decreases in body weight (5-10%) are needed to clinically improve CAD risk factors. Our data suggested that a 10% reduction in body weight is as effective in improving the metabolic profile as a 20% decrease in body weight. Thus, the question are : " Is it possible to further improve the metabolic profile over that 5-10% weight loss threshold?" and "Could several 5-10% body weight loss (intermittent weight loss approach) have additive effects on the metabolic profile?". We would like to follow-up on these observation to better understand 1) the association between weight loss and improvements in the metabolic profile and 2) why minor decreases in body composition and body fat distribution are as effective as more important reduction.

ELIGIBILITY:
Inclusion Criteria:

* Women who had stopped menstruating for more than 1 year
* Waist circumference > 90 cm
* Sedentary (< 2 times a week of structured exercise)
* Non-smokers
* Low to moderate alcohol consumers (< 2 drinks per day).

Exclusion Criteria:

* We excluded subjects with the following conditions based on medical history and physical examination and on laboratory testing of kidney and liver functions, serum TSH, fasting glucose and lipid profile, and 75g-OGTT
* Cardiovascular disease, peripheral vascular disease or stroke
* Diabetes
* Moderate to severe hypertension (resting blood pressure > 170/100 mm Hg);
* Body weight fluctuation > 5 kg in the previous 6 months
* Thyroid or pituitary disease
* Hormonal replacement therapy at any time during the previous 6 months
* Medication that could affect the metabolic profile

Ages: 51 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-09; Study Completion 2007-06

PRIMARY OUTCOMES:
Body composition (fat mass and lean body mass): after 0, 5, 10, 15, 20 and 25 weeks, as well as 12-month post-intervention

SECONDARY OUTCOMES:
Fasting lipids: baseline, 5, 10, 15, 20 and 25 weeks, as well as 12-month post-intervention
Resting metabolic rate: baseline, 5, 10, 15, 20 and 25 weeks, as well as 12-month post-intervention
Resting blood pressure: baseline, 5, 10, 15, 20 and 25 weeks, as well as 12-month post-intervention
OGTT: baseline and 25 weeks
Dietary habits: baseline,25 weeks and 12-month post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Martin Brochu, PhD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Institut universitaire de gériatrie de Sherbrooke, Sherbrooke, Quebec, Canada